CLINICAL TRIAL: NCT01122706
Title: Efficacy of Taiji Training as a Program for Stress Prevention - a Randomized, Waiting List Controlled Longitudinal Study With Healthy Subjects
Brief Title: Efficacy of Taiji Training as a Program for Stress Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Nedeljkovic Marko / MSc, University of Bern, Institute of Complementary Medicine KIKOM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 058/10
Record Dates: First submitted 2010-04-12; First posted 2010-05-13 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Primary Prevention; Stress; Tai ji; Adult
Keywords: tai ji; psychosocial stress; primary prevention; Trier Social Stress Test; salivary cortisol; salivary alpha amylase; heart rate variability; stress management
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taiji (Experimental): 35 healthy participants will regularly during 12 weeks attend Taiji training classes twice a week for one hour. (Sept. 6th till Nov. 25th 2010).
  Interventions: Other: Taiji training
- waiting list control group (No Intervention): 35 healthy participants are not allowed to attend any Taiji training during the intervention period (Sept. 6th till Nov. 25th 2010).

INTERVENTIONS:
Other: Taiji training — Taiji training during 12 weeks (twice a week for 1 hour) (Sept. 6th till Nov. 25th 2010). The first 18 sequences of a series of 37 movements of the short form Yang style Taiji will be taught. The focus will be on memorizing the series of movements, developing a regular training routine and working on body alignment and flow of the movements.
  Other Names: Taiji; Tai Chi; Tai Chi Chuan; Taijiquan
  Arms: Taiji

SUMMARY:
Background: Excessive exposure to psychosocial stress can be a potent trigger for somatic diseases and psychological disorders, a cause for missing work, and eventually lead to high economic loss. Therefore, for health and economic reasons the assessment of effectiveness of stress preventive interventions is of high relevance. According to several clinical studies, Taiji, a Chinese form of mindful and gentle movements, can significantly reduce symptoms of somatic diseases and psychological disorders. Some recently conducted Taiji-studies with healthy subjects indicate a stress protective effect. However, the stress protective impact of Taiji regarding psychosocial stress has not yet been examined.

Objective: To investigate the efficacy of a 12 week Taiji training as a stress prevention program by measuring psychosocial stress reactivity in a laboratory setting, as well as the subjective perception of stress and coping-resources in daily life of 70 healthy volunteers.

Hypothesis: Healthy subjects attending a 12 week Taiji course (frequency: twice a week for 1h) will show significantly reduced psychobiological reactivity, decreased stress perception and increased coping-resources on a standardized psychosocial stress test compared with healthy subject of the waiting list.

DETAILED DESCRIPTION:
Background:

Excessive exposure to psychosocial stress can be a potent trigger for somatic diseases and psychological disorders, a cause for missing work, and eventually lead to high economic loss. Therefore, for health and economic reasons the assessment of effectiveness of stress preventive interventions is of high relevance. According to several clinical studies, Taiji, a Chinese form of mindful and gentle movements, can significantly reduce symptoms of somatic diseases and psychological disorders. Some recent Taiji-studies with healthy subjects indicate a stress protective effect. However, since these findings mainly focus on effects during or immediately after a Taiji training session, their study designs and outcome measures are not comparable with existing stress prevention efficacy studies and their sample sizes are generally too small, the present available results remain inconclusive. Also, the impact of a Taiji training on psychosocial stress has not been assessed so far.

Objective:

The objective of this study is to assess the efficacy of a 12 week Taiji training as a stress prevention program by measuring psychosocial stress reactivity in a laboratory setting, subjective perception of stress and coping-resources of 70 healthy subjects in daily life.

Methods:

The Trier Social Stress Test (TSST) will be used to measure the psychobiological stress reactivity. Salivary cortisol, alpha amylase, heart rate and heart rate variability will be measured in each subject to asses stress reactivity, Also, the primary appraisal secondary appraisal (PASA) questionnaire and the multidimensional mood questionnaire (MDBF) will be used to assess psychological stress reactivity, and a visual analogue scale (VAS) to measure perceived stressfulness.

Additionally to the TSST setting, pre-, post-intervention and 2 months follow up measurements will be taken. The following tools will be used: Perceived Stress Scale (PSS), Stress Reactivity Scale (SRS)(to assess perceived stress), and self-efficacy-expectancy questionnaire (SWE), questionnaire for measuring wellbeing (FEW-16), Freiburg mindfulness inventory (FMI) and self compassion scale (SCS) (to assess perceived coping resources).

ELIGIBILITY:
Inclusion Criteria:

* ready to participate in the Taiji-intervention group as well as in the Waiting list control group
* mentally healthy
* physically healthy
* fluent in German (written and spoken)

Exclusion Criteria

* previous practical experience with Taiji-exercises
* previous practical experience with the Trier Social Stress Test
* being absent for more than one week between Sept. 6th and Nov. 25th 2010
* daily alcohol consumption more than two alcoholic drinks
* daily tobacco consumption more than five cigarettes per day
* any kind of drug consumption
* pregnancy
* intake of hormonal compounds i.e. birth control pill and hormon replacement therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) with respect to increase of salivary cortisol titer | durring the Trier Social Stress Test
  saliva samples will be taken 8 times during the Trier Social Stresstest. Salivary cortisol reactivity in response to this psychosocial stress test will be calculated by aggregating cortisol data of all 8 saliva samples in an AUC value with respect to increase.

SECONDARY OUTCOMES:
salivary alpha amylase reactivity to psychosocial stress | 8 times during the Trier Social Stress Test (which lasts 2h)
heart rate | continuously during the Trier Social Stress Test (which lasts 2h)
heart rate variability | continuously during the Trier Social Stress Test (which lasts 2h)
perceived stress | before, after the Taiji training and 2 months follow up
  to be measured by using the percieved stress scale (PSS)
self-efficacy-expectancy | before, after the Taiji training and 2 months follow up
  to be measured by using the self-efficacy-expectancy questionnaire (SWE)
wellbeing | before, after the Taiji training and 2 months follow up
  to be measured by using the questionnaire for measuring wellbeing (FEW-16)
Mindfulness | before, after the Taiji training and 2 months follow up
  to be measured by using the Freiburg mindfulness inventory (FMI)
Self Compassion | before, after the Taiji training and 2 months follow up
  to be measured by using the self compassion scale (SCS)

CONTACTS AND LOCATIONS:
Overall Officials: Marko Nedeljkovic, MSc, Principal Investigator — Institute of Complementary Medicine KIKOM
Locations (1):
- University of Bern, Institute of Complementary Medicine KIKOM, Bern, Switzerland

REFERENCES:
- [Background] Figueredo VM. The time has come for physicians to take notice: the impact of psychosocial stressors on the heart. Am J Med. 2009 Aug;122(8):704-12. doi: 10.1016/j.amjmed.2009.05.001. PMID 19635269
- [Background] Raison CL, Miller AH. When not enough is too much: the role of insufficient glucocorticoid signaling in the pathophysiology of stress-related disorders. Am J Psychiatry. 2003 Sep;160(9):1554-65. doi: 10.1176/appi.ajp.160.9.1554. PMID 12944327
- [Background] Klein PJ, Adams WD. Comprehensive therapeutic benefits of Taiji: a critical review. Am J Phys Med Rehabil. 2004 Sep;83(9):735-45. doi: 10.1097/01.phm.0000137317.98890.74. PMID 15314540
- [Background] Esch T, Duckstein J, Welke J, Braun V. Mind/body techniques for physiological and psychological stress reduction: stress management via Tai Chi training - a pilot study. Med Sci Monit. 2007 Nov;13(11):CR488-497. PMID 17968296
- [Background] Dickerson SS, Kemeny ME. Acute stressors and cortisol responses: a theoretical integration and synthesis of laboratory research. Psychol Bull. 2004 May;130(3):355-91. doi: 10.1037/0033-2909.130.3.355. PMID 15122924
- [Derived] Nedeljkovic M, Ausfeld-Hafter B, Streitberger K, Seiler R, Wirtz PH. Taiji practice attenuates psychobiological stress reactivity--a randomized controlled trial in healthy subjects. Psychoneuroendocrinology. 2012 Aug;37(8):1171-80. doi: 10.1016/j.psyneuen.2011.12.007. Epub 2012 Jan 4. PMID 22222120